CLINICAL TRIAL: NCT06774989
Title: Real-life Pharmacological Monitoring of Encorafenib-Binimetinib in the Treatment of Metastatic Melanoma
Acronym: SPEBINI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240895; 2024-A00842-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-12-03; First posted 2025-01-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Melanoma (Skin)
Keywords: melanoma; targeted therapy; BRAF and MEK inhibitors; pharmacokinetics
MeSH Terms: conditions — Melanoma; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, the prognosis for BRAFV600E-mutant metastatic melanoma has been transformed with targeted therapies combining BRAF and MEK inhibitors (dabrafenib-trametinib and encorafenib-cobimetinib), which have improved progression-free survival and overall survival. However, adverse events are very frequent, and a significant proportion of patients progress secondarily. Several clinical studies have shown that inter-individual variability in plasma exposure to BRAF inhibitors (dabrafenib, vemurafenib) or MEK inhibitors (trametinib) may contribute in part to the occurrence of severe toxicities, and on the efficiency of the treatment. To our knowledge, no data are currently available on the exposure/toxicity relationship for encorafenib and binimetinib.

The aim of this study is to assess the association between plasma exposure of encorafenib and binimetinib and the occurrence of dose-limiting toxicity during the first 3 months of treatment.

Our secondary objectives are the identification of factors of variability in plasma exposure to encorafenib and binimetinib, the assessment of the exposure-response relationship to treatment (PFS, OS), the evaluation of the influence of the residual plasma concentration of checkpoint inhibiting antibodies (nivolumab, pembrolizumab, ipilimumab) in the first month on the occurrence of dose-limiting toxicity during treatment with encorafenib/binimetinib. Also, the investigators will study the relationship between the kinetics of circulating tumour DNA levels and plasma exposure to encorafenib and binimetinib. Finally, the investigators will assess compliance with treatment.

All patients over the age of 18 receiving encorafenib-binimetib for BRAF-mutated metastatic or locally advanced non-operable melanoma, regardless of line, in our 5 centres, will be included.

After the patient has been informed and informed that he or she does not wish to be included in the study, an additional blood test will be taken during follow-up visits to the HDJ or specific follow-up consultation for his or her metastatic melanoma, where blood sampling is already planned as part of the treatment, during 1 year.

The tubes will be sent to the laboratories for analysis in the usual way as part of routine care. A self-questionnaire will be given to the patient at different follow-up visits.

Research data, including clinical, biological and self-questionnaire data, will be collected in the study via a web interface (e-CRF).

Follow-up of the population will follow the rhythm of visits scheduled as part of the usual care of patients with melanoma undergoing targeted therapy. the investigators plan a 1-year sampling period, and a 2-year clinical follow-up period for each patient from the time of inclusion. Finally, the investigators plan a period of 1 year to analyze the data and write the article.

Statistical analysis will be carried out by the investigating team (R software).

DETAILED DESCRIPTION:
Our study focuses on adult patients with BRAFV600-mutant metastatic melanoma treated with encorafenib and binimetinib, or encorafenib alone (regardless of treatment line). Encorafenib and binimetinib are BRAF and MEK inhibitors, respectively. They constitute a combination of oral targeted therapies, with marketing authorization since 2018 in metastatic melanoma in patients with BRAFV600-mutated melanoma, in first-line treatment or after progression on immunotherapy.

It is taken orally, at an initial dose of :

* 450 mg (six 75 mg capsules) once daily for encorafenib ;
* 45 mg (3 x 15 mg tablets) twice daily, 12 hours apart, for a total daily dose of 90 mg.

  5 recruiting centers (APHP): Hôpital Ambroise Paré (Boulogne-Billancourt), Hôpital Avicenne (Bobigny), Hôpital Cochin (Paris 14), Hôpital Henri Mondor (Créteil) and Hôpital Bichat (Paris 18).

For the purposes of this research, subjects will be identified as follows:

center no. (3 numeric positions) - person selection order no. in center (4 numeric positions) - initial surname - initial first name This reference is unique and will be kept for the duration of the research.

Patients will be recruited from the dermatology departments of 5 recruiting centers.The investigator, a dermatologist, will inform the patient at the time of his or her usual follow-up in the context of melanoma care. Notice of participation in the research will be collected and transcribed into the patient's medical record. The present protocol does not interfere with patients' medical management of their melanoma-related pathology. Eligible patients will be invited to take part in the study by the investigating physician during a follow-up visit in HDJ or a specific follow-up consultation for their melanoma. During the visit, the investigating physician will inform eligible patients about the study and answer any questions they may have about its purpose, constraints, foreseeable risks and expected benefits. After reading the information letter and taking some time to think about it, the doctor will obtain the patient's opinion from and an additional 20 ml blood sample will be taken. Temporality :

* Determination of plasma concentrations of immune checkpoint inhibitor antibodies: D0 and M1 if treated with checkpoint inhibitors within the last 6 months (pembrolizumab, nivolumab, ipilimumab).
* Measurement of encorafenib-binimetinib plasma concentrations: M1, M2, M4 or M1, M3 of combotherapy initiation, depending on the center, then after 6 months of treatment every 2 to 3 months and at the time of progression (if not on the day of a re-evaluation HDJ when sampling is already planned) or of a severe toxic episode for which the patient consults, for 1 year. NB: The patient can be sampled at any time between two doses. Encorafenib must be taken in the evening (to avoid skipping doses on the morning of sampling).
* Essential information on the sampling sheet: dose, date and time of last dose for each drug, date and time of sampling.
* Detection of circulating tumor DNA: D0, M1, M2 then every 2 or 3 months for 1 year, only if performed as part of routine care

Sampling and transport methods:

* Determination of checkpoint inhibitor antibody concentrations: 1 x 5ml tube sent to UF Biologie du Médicament-Toxicologie at Cochin for all centers except Bichat (sent to Saint Louis)
* Determination of encorafenib-binimetinib concentrations :
* for patients at Ambroise-Paré hospital: 1 x 5 ml tube sent to the pharmacology laboratory at Raymond Poincaré hospital (Pr JC Alvarez)
* for patients at Hôpital Bichat: 1 x 5 ml tube sent to the pharmacology laboratory at Hôpital Saint Louis.
* for patients from the 3 other centers: 1 x 5 ml tube sent to the UF Biologie du Médicament-Toxicologie at Hôpital Cochin.
* Detection of circulating tumor DNA (only if performed as part of routine care) :
* for patients at Ambroise-Paré Hospital: 1 x 10-ml EDTA tube sent to Pr Jean-François Emile in molecular biology at Ambroise-Paré Hospital
* for patients at Avicenne Hospital: 1 x 10 ml EDTA tube sent to Pr Schischmanoff and Dr Fabre in molecular biology at Avicenne Hospital
* for patients at Hôpital Bichat: 1 x 10 ml EDTA tube sent to Pr ANNE COUVELARD in molecular biology at Hôpital Bichat.
* for patients from the 2 other centers (Hôpital Cochin and Hôpital Mondor): 1 x 5 ml cell-free DNA tube sent to the anatomopathology and molecular biology laboratory at Hôpital Européen Georges Pompidou.

Essential information on the sampling sheet: dose, date and time of last dose for each drug, date and time of sampling.

Dosage methods :

* Determination of plasma drug concentrations by liquid chromatography-mass spectrometry (LC-MS/MS)
* Detection of circulating tumor DNA (BRAFV600 allele) in peripheral blood by digital droplet PCR (15)

Dosing centers :

* Pharmacology laboratories (drug dosage) :

  * Hôpital Cochin and Hôpital Saint Louis: encorafenib, binimetinib, pembrolizumab, nivolumab, ipilimumab
  * Raymond Poincaré Hospital: encorafenib, binimetinib
* Pathology and molecular biology laboratories (detection of circulating tumor DNA):

  * Ambroise Paré Hospital
  * Georges Pompidou European Hospital
  * Bichat Hospital Tubes transferred by sorting centers according to standard procedure. Bayesian estimation of residual concentrations (Cmin ) and total exposure (AUC) between two intakes using a KP/POP model.

To this end, the investigators will build two population pharmacokinetic models to explore the factors of variability in the pharmacokinetics of encorafenib and binimetinib. Based on these models, residual concentrations of each molecule will be estimated to explore the PK/PD relationship of encorafenib and binimetinib. The methodology used to build the models will be based on recommendations in the literature (16) At the end of the research, the samples will be destroyed. Follow-up of the population will follow the rhythm of visits scheduled as part of the usual care of patients with melanoma undergoing targeted therapy. the investigators plan a sampling period of 1 year, and a clinical follow-up period of 2 years for each patient from inclusion. Finally, the investigators plan a 1-year period for data analysis and article writing Clinical and biological data are collected at each visit for 2 years. An additional 20-ml blood sample (3 tubes with EDTA) is taken in the first year. Sampling and transport procedures are identical to those for the inclusion visit.

Non-interventional research involving the human body poses no risk to patients. Adverse reactions observed in patients taking part in research are reported by investigators in accordance with local vigilance plans set up as part of their care activities.

The data corresponding to the various clinical and biological examinations will be completed by Dr Sarah Bouchereau in the RedCap database from the medical record and the analysis results retrieved from the laboratories.

Questionnaire data will be entered directly into the RedCap database by Dr Bouchereau.

Patient anonymity will be ensured, in accordance with the AP-HP promoter's procedure, by a reference in the form of a center code (3 digits), a center inclusion number (4 digits) and the initials (one letter for the surname and one letter for the first name) of the person taking part in the research on all documents required for the research.

Access to e-CRF via the Internet will be secured by a username and password, and data flow will be encrypted using the https protocol.

Clinical data from each center will be collected in order to gather the following data from medical records (CRH, CR de consultation) sent to Pr Elisa Funck-Brentano, Dr Sarah Bouchereau and Benoit Blanchet.

The data will be recorded by each investigator in the patient's file during the usual follow-up consultations. Sarah Bouchereau, Elisa Funck-Brentano and Benoit Blanchet, who will have been notified of each letter (via ORBIS, mssanté secure messaging system), will then transfer these data, which will be considered as source data, directly into the RED Cap anonymized e-CRFs.

Self-questionnaires completed by patients will be kept in the study binder.

In accordance with GCP :

* the sponsor is responsible for obtaining the agreement of all parties involved in the research to guarantee direct access to all research sites, source data, source documents and reports for quality control and audit purposes by the sponsor,
* investigators will make available to those responsible for monitoring and quality control, in the event of an audit of research involving the human person, the documents and individual data strictly necessary for this control, in accordance with the legislative and regulatory provisions in force Source documents, defined as any original document or object that can be used to prove the existence or accuracy of data or facts recorded during the course of research, will be kept for 15 years by the investigator, or by the hospital in the case of hospital medical records.

Those responsible for quality control in research involving the human body (article L.1121-3 of the French Public Health Code), will take all necessary precautions to ensure the confidentiality of information relating to the research, to the persons involved, and in particular to their identity, and to the results obtained.

These people, like the investigators themselves, are bound by professional secrecy.

During and at the end of research involving the human person, data collected on subjects and transmitted to the sponsor by the investigators (or any other specialist) will be rendered non-identifying.

Under no circumstances may the names or addresses of the persons concerned appear in plain text.

Only the initials of the surname and first name will be recorded, together with a coded number specific to the research indicating the order of inclusion of subjects.

The sponsor will ensure that each person taking part in the research has given his or her consent for access to individual data concerning him or her and strictly necessary for the quality control of the research.

Identification of the person in charge and the location of data entry and processing management Sarah Bouchereau will enter the non-identifying data of all patients on a CRF-type paper medium, then transfer it to an Excel-type digital data collection table.

Statistical analysis will be carried out by the investigating team. Based on data from the Columbus Phase 3 trial (14)the rate of discontinuation due to toxicity was 6% in the (encorafenib/binimetinib) arm, and 48% of patients had their dose reduced.

Given that DLT (treatment discontinuation or dose reduction) is our primary endpoint, the investigators considered a frequency of DLT occurrence of 50% in our study.

Furthermore, the investigators hypothesize that the 25% of patients with the highest encorafenib exposure (quartile 4, Q4) will more frequently present with DLT than patients with plasma exposures within Q1-Q3 (80% vs. 40%, respectively). Thus, with a two-sided α-risk of 5% and power of 80%, 59 patients will need to be included in the study to confirm our hypothesis. the investigators therefore plan to include 66 patients in order to take into account 10% of potential los de vus.

Population analyzed: all patients meeting inclusion and exclusion criteria will be analyzed

Rules for handling missing data: missing data will not be taken into account.

Definitions :

* Dose-limiting toxicity: occurrence of toxicity requiring discontinuation of encorafenib and/or binimetinib AND/OR reduction in dose by one dose level within the first 6 months of treatment .
* Progression-free survival (PFS) will be calculated from the date of D1 of encorafenib/binimetinib to the date of diagnosis of progression (according to RECIST criteria) 16 or the date of last news if the date of progression is unknown .
* Overall survival (OS) will be calculated from the date of D1 of encorafenib/binimetinib until the date of death or the date of last news if the date of death is not known.

General statistical approach for exposure-response analysis :

* Descriptive study of primary endpoints
* Group comparison (Q1-3 vs Q4) with Chi2 or Fisher test for qualitative variables and Wilcoxon test for quantitative values.
* Logistic regression for factors predictive (including AUC and Cmin for each molecule) of the occurrence of dose-limiting toxicity. Factors associated with the occurrence of dose-limiting toxicity with a p-value < 0.1 in univariate analysis will be included in a multivariate model.
* Cox model for prognostic factors (including mean AUC and Cmin over the first 3 months for each molecule) for PFS and OS. Factors associated with progression or death with a p-value < 0.1 in univariate analysis will be included in a multivariate model.

The aim is to have no missing data for the main evaluation criterion. For other variables, missing data may be determined by imputation if their proportion does not exceed 10%.

Data quality control for statistical analyses consists in checking that the data in the observation books are complete, consistent and plausible. In the event of an anomaly, the investigator will be asked to correct it. If a verification is necessary in a source document, it can only be carried out by a member of the medical team supervising the subject.

The information notes, including the record of non-opposition, will be kept by the head of the medical team supervising the subjects for a period of 15 years.

Only the initials of the surname and first name will be recorded, along with a coded number specific to the search.

The sponsor will ensure that each person taking part in the research has not objected to access to individual data concerning him or her and strictly necessary for the quality control of the research.

In accordance with article L1121-1-1 of the French Public Health Code, no non-interventional research may be carried out on a person who has objected to it after having been provided with the information required under article L11222-1 of the same code.

The patient is allowed a 15-day cooling-off period, no later than the day before the inclusion visit, between the time he or she is informed and the time the investigator signs the no-objection form. The information note is given at the screening visit.

In urgent cases, when the introduction of encorafenib and binimetinib treatment cannot be delayed, this delay can be reduced to 2 hours in order to be able to include the patient. This study should in no way delay treatment.

Patient information will be provided orally by the dermatologist investigator during follow-up visits for metastatic melanoma, who will give the patient an information document. The patient's information and non-opposition will be documented in the patient's medical record.

A copy of the information document is given to the person prior to participation in the research.

The information given to the subject will be recorded in his or her medical file.

The non-opposition of the subject will be recorded in his medical file by the investigator or the qualified person who collects it.

ELIGIBILITY:
Inclusion Criteria:

Adults ≥ 18 years of age

* Histologically confirmed advanced melanoma, stage III/stage IV inoperable (primary cutaneous, mucosal or unknown)
* Treatment with encorafenib and/or binimetinib, whatever the line of treatment, for curative purposes.
* Affiliated to a social security scheme or beneficiary of such a scheme
* informed and non-opposition collected.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with BRAFV600-mutated metastatic melanoma treated with encorafenib and binimetinib (any line of therapy).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
association between the plasma exposure of encorafenib and binimetinib and the occurrence of dose-limiting toxicity | 3 months
  association between the plasma exposure of encorafenib and binimetinib and the occurrence of dose-limiting toxicity during the first 3 months of treatment

SECONDARY OUTCOMES:
plasma exposure to encorafenib | Month 1, Month 2, Month 6, Month 9 and 1 year
  therapeutic compliance will be assessed both by the physician during follow-up consultations and by a standardized questionnaire (GIRERD questionnaire) filled in by the patient during follow-up consultations (M1, M2 then every 2 or 3 months for 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa FUNCK-BRETANO, MD, PhD, Principal Investigator — Department of Oncology-Dermatology, Ambroise Paré Hospital - APHP
Locations (1):
- Department of Oncology-Dermatology, Ambroise Paré Hospital - APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: Undecided